CLINICAL TRIAL: NCT02258412
Title: Evaluation of Antimicrobial Efficacy of Two Hand Hygiene Products in ICUs Using Hand Prints
Brief Title: Evaluation of Two Hand Hygiene Products in ICUs
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Solventum US LLC (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EM-05-013218
Record Dates: First submitted 2014-09-17; First posted 2014-10-07 (Estimated); Results first posted 2017-05-16 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-09

CONDITIONS: Hand Hygiene Effectiveness
Keywords: antimicrobial; efficacy; hand; hygiene; bacteria
MeSH Terms: interventions — Hand Sanitizers; Chromogranins; Ethanol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Alcohol hand sanitizer foam (Active Comparator): Alcohol foam hand sanitizer applied with 1 pump into hands, spread over hands up to the wrist and rubbed until dry. Foam will be applied twice approximately 15-30 minutes apart on one day.
  Interventions: Drug: Alcohol hand sanitizer foam
- hand antiseptic with CHG and alcohol (Active Comparator): Hand antiseptic is applied by dispensing 1 pump into hands, spreading over the hands up to the wrist, and rubbing until dry. Hand antiseptic will be used twice approximately 15-30 minutes apart on one day.
  Interventions: Drug: hand antiseptic with CHG and alcohol

INTERVENTIONS:
Drug: hand antiseptic with CHG and alcohol — HCWs will be randomized to use one product on one day and the other product on another day at least 3 days apart. Each product will be applied using 1 pump from its dispenser and rubbed over the hands until dry. Gloves will be worn while the HCW is in the patient room. Upon exit from the room, HCW will washoout with that same product. One imprint will be made of the non-dominant hand onto media containing neutralizers. That hand will be gloved with a white cotton glove. The HCW will work in the common areas with timing recorded. Upon leaving the common area, the dominant ungloved hand will be imprinted onto a fresh media plate containing neutralizers.
  Other Names: Avagard CHG Hand Antiseptic with Moisturizers; Purell Advanced Instant Hand Sanitizer Foam
  Arms: hand antiseptic with CHG and alcohol
Drug: Alcohol hand sanitizer foam — Alcohol foam hand sanitizer applied with 1 pump into hands, spread over hands up to the wrist and rubbed until dry. Foam will be applied twice approximately 15-30 minutes apart on one day
  Other Names: Purell Instant Sanitizer Foam
  Arms: Alcohol hand sanitizer foam

SUMMARY:
This study will evaluate the immediate antimicrobial efficacy and persistence of two hand hygiene products on ICU Health Care Worker's skin flora by measuring bacterial organisms on hands using the hand print method. It is hypothesized that the product containing Chlorhexidine gluconate will provide more persistence than the alcohol product, resulting in less bacterial growth on the hand print plates. In addition, environmental monitoring for cleanliness will be captured from high touch surfaces in ICU patient rooms and common areas using Rodac plates and adenosine triphosphate tests.

DETAILED DESCRIPTION:
Crossover study with 50 Health care workers using each product with a minimum of 3 days in between. Products will be applied twice as per manufacturer's instructions for a Healthcare Personnel Handwash followed by immediate hand print. Persistent hand prints will be collected after exposure to environmental contaminants in the common areas. Hand prints will also be collected from one hand of 60 patients cared for by a participating Health Care Worker and gloved hand of Health Care Worker. All media contain neutralizers to inactivate active ingredients in each product and on surfaces. Each hand print plate's area of growth will be measured for Colony Forming Units using computerized software.

ELIGIBILITY:
Inclusion Criteria:

* HCW willing to participate in the study
* HCW willing to use non-Triclosan soap when soap is necessary throughout the study
* HCW who will don gloves prior to ICU patient room entry

Exclusion Criteria:

* Use of any CHG -containing products ( liquid hand soap, Sage wipes) on the ICU 72 hours prior to study initiation and throughout study
* HCW with patient bandage or other dressing on palm(s)
* Known sensitivity or allergy to CHG or alcohols in hand hygiene products
* Known sensitivity or allergy to the following components: Lecithin, Polysorbate 80,Trypticase Soy Agar, sodium bisulfate, sodium thioglycollate, sodium thiosulfate
* History of skin allergies

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-10; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abhishek Deshpande, MD, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Deshpande A, Fox J, Wong KK, Cadnum JL, Sankar T, Jencson A, Schramm S, Fraser TG, Donskey CJ, Gordon S. Comparative Antimicrobial Efficacy of Two Hand Sanitizers in Intensive Care Units Common Areas: A Randomized, Controlled Trial. Infect Control Hosp Epidemiol. 2018 Mar;39(3):267-271. doi: 10.1017/ice.2017.293. Epub 2018 Jan 31. PMID 29382400

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place from October 2014-January 2015 at 3 MICUs within the same hospital
Pre-assignment Details: Subjects were enrolled on the same day as treatment; subjects were required to meet inclusion/exclusion criteria to qualify for enrollment
Groups:
- Alcohol + CHG First: Healthcare workers who received product with alcohol + CHG prior to product with alcohol only
- Alcohol Only First: Healthcare workers who received product with alcohol only prior to product with alcohol + CHG
- Patient: Patients received no treatment, but were cared for by healthcare workers who enrolled in the study
Period: Overall Study
Arm/Group | Alcohol + CHG First | Alcohol Only First | Patient
Started | 26 | 25 | 61
Completed | 26 | 25 | 61
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alcohol + CHG First | Alcohol Only First | Patient | Total
Number analyzed (Participants) | 26 | 25 | 61 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | NA (NA) — Subject age was not recorded as it is not relevant to the study outcome | NA (NA) — Subject age was not recorded as it is not relevant to the study outcome | NA (NA) — Subject age was not recorded as it is not relevant to the study outcome | NA (NA) — Subject age was not recorded as it is not relevant to the study outcome
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — Subject gender was not recorded as it is not relevant to the study outcome | NA — Subject gender was not recorded as it is not relevant to the study outcome | NA — Subject gender was not recorded as it is not relevant to the study outcome | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | NA — Subject gender was not recorded as it is not relevant to the study outcome | NA — Subject gender was not recorded as it is not relevant to the study outcome | NA — Subject gender was not recorded as it is not relevant to the study outcome | NA — Total not calculated because data are not available (NA) in one or more arms.
Region of Enrollment [Number; unit: participants]
  United States | 26 | 25 | 61 | 112

OUTCOME MEASURES:

1. Primary Outcome: Bacterial Colony Forming Units Present on Hand Prints After Time Spent in Common Areas
Description: Hand print plates will be collected from HCWs immediately after use of hand hygiene product and after time spent in common areas. Each HCW will use both products at least 3 days apart. Hand print plates from each product for each HCW will be compared.
Time Frame: On each of 2 days, Hand print plates collected from one hand immediately after product use (T0) and from other hand after time spent in MICU common areas
Measure: Mean (95% Confidence Interval); unit: log(10) transformed CFU
Arm/Group | Alcohol Hand Sanitizer Foam | Hand Antiseptic With CHG and Alcohol
Number analyzed (Participants) | 51 | 51
log(10) transformed CFU | 2.17 [2.07 to 2.27] | 1.81 [1.67 to 1.95]

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Alcohol + CHG First | Alcohol Only First | Patient
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/25 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/25 | 0/61
Other Adverse Events (participants affected / at risk) | 0/26 | 0/25 | 0/61

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less